CLINICAL TRIAL: NCT04518345
Title: A Phase 1b/2 Study of TP-0903 in Patients With Acute Myeloid Leukemia and FLT3 Mutations
Brief Title: TP-0903 for the Treatment of FLT3 Mutated Acute Myeloid Leukemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Uma Borate (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19229; NCI-2020-04292 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-30; First posted 2020-08-19 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; dubermatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dubermatinib) (Experimental): FLT3 AML WITH RELAPSED/REFRACTORY DISEASE:
  INDUCTION: Patients receive dubermatinib PO QD on days 1-21. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients with clinical or hematologic response and not transplant eligible may continue dubermatinib until loss of response/clinical benefit. Patients with clinical or hematologic response and transplant eligible may continue dubermatinib until one week prior to admission.
  Interventions: Drug: Azacitidine; Drug: Dubermatinib

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Dubermatinib — Given PO
  Other Names: TP 0903; TP-0903; TP0903

SUMMARY:
This phase IB/II trial studies the best dose of TP-0903 and how well it works when given alone or with azacitidine in treating patients with FLT3 gene mutated acute myeloid leukemia. TP-0903 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving TP-0903 alone or with azacitidine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a tolerable dose of dubermatinib (TP-0903) monotherapy for relapsed/refractory patients with FLT3 acute myeloid leukemia (AML).

II. To determine the maximum tolerated dose (MTD) of TP-0903 with azacitidine in untreated unfit patients with FLT3 AML.

III. To determine the complete remission (CR) or complete remission with partial hematologic recovery (CRh) rate following induction therapy with TP-0903 in relapsed/refractory patients or TP-0903 with azacitidine therapy in untreated unfit patients with FLT3 AML.

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of TP-0903 as a single agent and in combination with or azacitidine.

II. To determine disease-free survival for patients achieving CR/CRh in each cohort.

III. To determine overall survival for patients in each cohort. IV. To determine the proportion of patients who go to transplant.

EXPLORATORY OBJECTIVES:

I. To conduct pharmacokinetic studies of TP-0903 alone and in combination with azacitidine.

II. To examine changes in circulating AXL, Gas6, FLT3 ligand, and other cytokines/chemokines by TP-0903.

III. To determine the impact of TP-0903 on the inhibition of kinase signaling (AXL, FLT3, STAT5, AURKA), and metabolomics in AML cells.

IV. To determine differentially expressed genes in bone marrow stromal cells and AML cells upon TP-0903 treatment.

V. To examine sensitivity and resistance patterns associated with TP-0903 by genomic, epigenomic, and transcriptomic profiling.

OUTLINE: This is a phase Ib, dose-escalation study of dubermatinib followed by a phase II study.

(FLT3 AML WITH RELAPSED/REFRACTORY DISEASE):

INDUCTION: Patients receive dubermatinib orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients with clinical or hematologic response and not transplant eligible may continue dubermatinib until loss of response/clinical benefit. Patients with clinical or hematologic response and transplant eligible may continue dubermatinib until one week prior to admission.

After completion of study treatment, patients are followed up followed every 3 months for up to 2 years from registration and then every 6 months for up to 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML and the presence of FLT3-ITD mutation
* Patients with secondary AML or therapy related disease (t-AML) are eligible
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0mg/dL unless due to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Creatinine (Cr) clearance > 50 mL/min by Cockcroft-Gault calculation
* New York Heart Association (NYHA) Congestive Heart Failure (CHF) class II or better
* Cardiac ejection fraction ≥40%
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Ability to understand and willingness to sign the written informed consent document
* Human immunodeficiency virus (HIV) infection without history of acquired immunodeficiency syndrome (AIDS) and sufficiently high CD4 cells (> 400/mm^3) and low HIV viral loads (< 30,000 copies/ml plasma) not requiring anti-HIV therapy are eligible

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Treatment with hydoxyurea is permitted during cycle 1 to maintain white blood cell (WBC) < 40,000/uL
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system (CNS) malignancy
* Major surgery within 2 weeks before day 1
* Uncontrolled active infection. Patients with infection requiring parenteral antibiotics are eligible if the infection is controlled
* Patients with significantly diseased or obstructed gastrointestinal tract
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 6 months prior to enrollment, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding are excluded from this study. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with advanced malignant solid tumors
* Patients who are not able to swallow capsules or tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of dubermatinib (TP-0903) | Up to 28 days
  Determine a tolerable dose of TP-0903 monotherapy for relapsed/refractory patients with FLT3 AML.
Composite complete response (CR) rate | Up to 5 years post registration
  Will calculate the composite CR rate (complete remission [CR]/complete remission with incomplete count recovery [CRh) defined according to the 2017 European LeukemiaNet Acute Myeloid Leukemia recommendation.
Composite CR rate with partial hematologic recovery (CRh) rate | through study completion, an average of 1 year
  Will calculate the composite CR rate (CR/CRh), defined according to the International Working Group criteria and assessed at the end of induction.

SECONDARY OUTCOMES:
Disease-free survival | From the date of first CR/CRh until the first date of relapse/progression or death from any cause, assessed up to 5 years post registration
  Will be summarized by the Kaplan-Meier method to determine disease-free survival for patients achieving complete response CR/CRh in each cohort of the study.
The Number of patients who proceed to transplant | Up to 5 years post registration
  The number of patients who got to transplant
Overall survival | From the treatment start date until the date of death from any cause or date last known alive, assessed up to 5 years post registration
  Will be summarized by the Kaplan-Meier method.
Maximum grade of each type of adverse event | Up to 5 years post registration
  Will be recorded for each patient and summarized.
Incidence of treatment-related adverse events | Up to 5 years post registration
  Treatment-related adverse events, defined as possibly, probably or definitely related to study treatment per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be summarized separately.
Tolerability of TP-0903 | Up to 5 years post registration
  Reasons for treatment discontinuation and number of TP-0903 cycles received will be summarized and used to assess tolerability.

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) pharmacokinetics (PK) | Up to 5 years post registration
  Initial analysis of plasma PK data will include standard compartmental and noncompartmental methods. Descriptive statistics including means, standard deviations, and frequencies will be computed for all variables. Relationships between continuous variables will be performed using standard linear correlation and linear regression. Relationships between PK parameters such as maximum concentration with response will be performed using standard t-tests or Wilcoxon rank sum tests and illustrated using boxplots or other graphical displays.
Area under the plasma concentration (AUC) pharmacokinetics (PK) | Up to 5 years post registration
  Initial analysis of plasma PK data will include standard compartmental and noncompartmental methods. Descriptive statistics including means, standard deviations, and frequencies will be computed for all variables. Relationships between continuous variables will be performed using standard linear correlation and linear regression. Relationships between PK parameters such as area under curve with response will be performed using standard t-tests or Wilcoxon rank sum tests and illustrated using boxplots or other graphical displays.
Changes in cytokines/chemokines | Up to 5 years post registration
  Differences in cytokines/chemokines will be evaluated using paired t-tests or Wilcoxon signed rank tests. Values will be log transformed as appropriate to reflect biologic plausibility. Cytokines/chemokines to be measured include: AXL, GAS6, FLT3 ligand, GM-CSF, IL-6, IL-8, RANTES, MIP-1α, MCP-1, sCD40L, EGF, VEGF
Effect of TP-0903 on inhibition of phospho-protein expression Effect of TP-0903 on inhibition of phospho-protein expression Effect of TP-0903 on inhibition of phospho-protein expression Impact of TP-0903 on kinase signaling | Up to 5 years post registration
  Percent inhibition of phospho-protein expression in AML cells. Phospho-proteins to be measured include: phospho-FLT3, phospho-STAT5, phospho-AURKA/B, phosho-AXL
Patterns of sensitivity and resistance | Up to 5 years post registration
  Mutational status in AML cells will be determined in samples at baseline and during treatment. Mutations in genes with single nucleotide changes and indels at variant allele frequency (VAF) >0.1 will be reported. Mutations with decreasing VAF represent sensitivity, and increasing VAF represent resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Uma Borate, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04518345/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04518345/ICF_001.pdf